CLINICAL TRIAL: NCT07241572
Title: Evaluation of Perioperative Myocardial Injury in Patients Undergoing Below-knee Lower Extremity Surgery With Peripheral Nerve Block
Brief Title: Evaluation of Perioperative Myocardial Injury in Patients Undergoing Below-Knee Lower Extremity Surgery
Status: Recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: E2-25-11354
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Myocardial Ischemia; Diabetes Complication
Keywords: myocardial injury; Troponın I; diabetic neuropaty; MINS
MeSH Terms: conditions — Myocardial Ischemia; Diabetes Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients undergoing elective below-knee lower extremity surgery: All patients undergoing below-knee lower extremity surgery will have their high-sensitive troponin I levels monitored preoperatively and at the 24th and 48th hours postoperatively.
  Intraoperatively, routine anesthetic monitoring (SpO2, blood pressure, ECG, apical heart rate) will be recorded. The presence and duration of intraoperative hypotension, the need for inotropic support, the total dose (if any), the presence and duration of tachycardia and bradycardia, the amount of fluid administered, urine output, and the duration of surgery will be recorded.
  Postoperative complications will be recorded. Patients will be followed up for 30 days through the hospital registry and telemedicine at the investigator's discretion, and will be questioned about potential major cardiac events (MACE).
  Interventions: Diagnostic Test: high sensitive Troponin I

INTERVENTIONS:
Diagnostic Test: high sensitive Troponin I — High sensitive Troponin I used to predict myocardial damage

SUMMARY:
The aim of this observational study was to detect myocardial damage by monitoring high-sensitive troponin I levels in patients undergoing below-knee extremity surgery with peripheral nerve block.

The primary question it aims to answer is:

How effective are peroperative high-sensitive troponin I levels in predicting myocardial damage?

High-sensitive troponin I levels will be monitored intraoperatively and at 24 and 48 hours postoperatively.

DETAILED DESCRIPTION:
Peripheral nerve blocks are becoming increasingly popular in foot and ankle surgery. Patients undergoing peripheral nerve blocks have advantages such as shorter hospital stays, better postoperative pain relief, lower costs, and less opioid use.

A review of current literature revealed that myocardial damage has not been investigated in patients scheduled for below-knee lower extremity surgery. Therefore, we aimed to detect myocardial damage by monitoring high-sensitive troponin I levels, which is considered the most sensitive and effective test according to AHA/ACC (American College of Cardiology and American Heart Association) guidelines at our hospital. The secondary aim of the study was to determine which parameters correlate with myocardial damage.

Preoperatively, the patient's hemogram, biochemistry, and hsTroponin I measurements, all of which were requested during the preparation phase, will be recorded.

During the operation, the type of anesthesia, the amount of local anesthetic and adjuvant medication used for peripheral nerve blockade will be recorded.

Intraoperatively, routine anesthetic monitoring (SpO2, blood pressure, ECG, heart rate), intraoperative presence and duration of hypotension, need for inotropic support, total dose (if any), presence and duration of tachycardia and bradycardia, fluid volume administered, urine output, and operation time will be recorded.

Postoperatively, all patients will be monitored in their ward or intensive care unit. Routine hemogram, biochemistry, and hsTroponin I measurements will be repeated at 24 and 48 hours, and the results will be noted. Postoperative complications will be recorded.

Patients will be followed up for 30 days through the hospital registry and telemedicine at the investigator's discretion, and will be questioned about potential major cardiac events (MACE).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients undergoing below-knee lower extremity surgery
* Patients with ASA classifications I, II, III, and IV
* Patients who have consented before the procedure
* Patients who are literate and able to give consent

Exclusion Criteria:

* Patients in whom regional anesthesia is contraindicated
* Patients who refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing below-knee lower extremity surgery under peripheral nerve blockade
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
High sensitive Troponin I | 01.09.2025-10.01.2026
  peroperative High sensitive Troponin I
High sensitive Troponin I | 01.09.2025-11.01.2026
  postoperative 24th hour High sensitive Troponin I
High sensitive Troponin I | 01.09.2025-12.01.2026
  postoperative 48th hour High sensitive Troponin I

SECONDARY OUTCOMES:
hemodynamic parameters 1 | 01.09.2025-10.01.2026
  intraoperative blood pressure (mmHg)
hemodynamic parameters 2 | 01.09.2025-10.01.2026
  intraoperative oxygen saturation (%)
hemodynamic parameters 3 | 01.09.2025-10.01.2026
  heart rate (/min)

OTHER OUTCOMES:
unexpected events | 01.09.2025-10.02.2026
  Sudden myocardial infarction occurring during the operation or within 1 month after the operation
unexpected events | 01.09.2025-11.02.2026
  Cerebrovascular accident occurring during the operation or within 1 month after the operation
unexpected events | 01.09.2025-12.02.2026
  rehospitalization during the operation and within 1 month after the operation
unexpected events | 01.09.2025-13.02.2026
  Death during surgery or within 1 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Harun Zengin, Principal Investigator — harunzengin71@gmail.com
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
general demographic information, contact information, work names

REFERENCES:
- [Result] Park J, Hyeon CW, Lee SH, Kim J, Kwon JH, Yang K, Min JJ, Lee JH, Lee SM, Yang JH, Song YB, Hahn JY, Choi JH, Choi SH, Kim K, Ahn J, Gwon HC. Mildly Elevated Cardiac Troponin below the 99th-Percentile Upper Reference Limit after Noncardiac Surgery. Korean Circ J. 2020 Oct;50(10):925-937. doi: 10.4070/kcj.2020.0088. Epub 2020 Jul 24. PMID 32812403
- [Result] Horr S, Reed G, Menon V. Troponin elevation after noncardiac surgery: Significance and management. Cleve Clin J Med. 2015 Sep;82(9):595-602. doi: 10.3949/ccjm.82a.15076. PMID 26366956
- [Result] Devereaux PJ, Szczeklik W. Myocardial injury after non-cardiac surgery: diagnosis and management. Eur Heart J. 2020 May 1;41(32):3083-3091. doi: 10.1093/eurheartj/ehz301. PMID 31095334